CLINICAL TRIAL: NCT06931626
Title: Study of NMS-03305293, a Non-Trapping PARP1-Specific PARP Inhibitor in Relapsed Small Cell Lung Cancer
Brief Title: Study of NMS-03305293 in Adult Patient With Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARPA-293-004
Record Dates: First submitted 2025-04-04; First posted 2025-04-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMS-03305293 and Temozolomide (Experimental): NMS-03305293 will be dosed orally on days 1-28 of each 28-day cycle, at 100 mg twice daily. Temozolomide will be dosed orally on days 1-5 of each 28-day cycle, at 150 mg/m^2, based on patients' body surface area.
  Interventions: Drug: NMS-03305293; Drug: Temozolomide

INTERVENTIONS:
Drug: NMS-03305293 — Route of administration: Oral
Drug: Temozolomide — Route of administration: Oral Commercially available Temozolomide

SUMMARY:
This is an open-label study of NMS-03305293 with Temozolomide (TMZ) in patients with Small Cell Lung Cancer (SCLC). The aim of this study is to determine the safety and tolerability, as well as to evaluate the anti-tumor efficacy and pharmacokinetics of NMS-03305293 in combination with TMZ.

ELIGIBILITY:
Inclusion Criteria -

* Histologically confirmed extensive-stage Small Cell Lung Cancer (SCLC); must have failed prior front-line platinum-based therapy including immune therapy with relapse within 6 months followed by failed tarlatamab therapy, if available and appropriate, and no more than 3 total prior lines of systemic therapy (therapy terminated due to toxicity or drug shortage, in the absence of Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 progression, will be considered part of the same line). Sponsor may opt to allow history of treatment free interval from front-line longer than 6 months .
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient must have progressed radiographically on or after their most recent line of anticancer therapy and have measurable disease as defined by RECIST v1.1 (radiologically measured by the Investigator).
* The interval from prior antitumor treatment should be at least 2 weeks or 5 half-lives, whichever longer.
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 Grade ≤ 1 or to the baseline laboratory values as defined in the protocol.
* Patients must use highly effective contraception or true abstinence.
* Ability to swallow capsules intact (without chewing, crushing, or opening).

Exclusion Criteria -

* Current enrollment in another interventional clinical trial.
* Current treatment with other anticancer agents or devices.
* Major surgery, other than surgery for recurrent SCLC, within 4 weeks prior to treatment start.
* Patients with prior wide-field radiotherapy (RT) affecting at least 20 percent of the bone marrow.
* Histologically transformed SCLC, i.e. tumors initially diagnosed as Non-Small Cell Lung Cancer (NSCLC) or mixed lung adenocarcinoma
* Known paraneoplastic syndrome uncontrolled or that required therapeutic changes (either new/acute or chronic) in the 14 days prior to study entry
* Use of full-dose anticoagulants unless the International Normalized Ratio (INR) or a Partial Thromboplastin Time (PTT) is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks before enrollment.
* Treatment with concomitant medications known to be sensitive substrates of CYP2D6 and CYP2C19 that cannot be replaced with another treatment.
* Treatment with systemic immune modulators such as corticosteroids at prednisone equivalent dose of > 10 mg/day, cyclosporine and tacrolimus or radiotherapy within 28 days before treatment start.
* Breast-feeding women or women planning to breast feed during the study or within 3 months after study treatment.
* Known hypersensitivity to any component of NMS-03305293 or Temozolomide (TMZ) drug formulations.
* Known active, life-threatening or clinically significant uncontrolled systemic infection (bacterial, fungal, viral including Human Immunodeficiency Virus [HIV] positivity or Hepatitis B Virus [HBV] or Hepatitis B Virus [HCV] infections) requiring systemic treatment; HIV or Acquired Immune Deficiency Syndrome (AIDS)-related illness are allowed as long as controlled more than 6 months to undetectable on anti-HIV medications.
* Patients with QT interval using Fridericia standard (QTcF) interval >450 milliseconds or with risk factors for torsade de pointes (e.g., uncontrolled heart failure, uncontrolled hypokalemia, history of prolonged QTc interval or family history of long QT syndrome). For patients receiving treatment with concomitant medications known to prolong the QTc interval, replacement with another treatment prior to enrollment is mandatory. If concomitant use of anti-emetics is considered essential for the care of the patients, follow instruction in this protocol
* Known active gastrointestinal disease (e.g., documented gastrointestinal ulcer, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes or structural issues or ulcer that would impact on drug absorption.
* Any of the following in the previous 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, active bleeding disorder and interstitial lung disease.
* History of long QT disorder or familial sudden death syndromes or related syndromes in the opinion of the Investigator.
* Currently active second malignancy, except for adequately treated basal or squamous cell skin cancer and/or cone biopsied or post curative intention in situ carcinoma of the cervix uteri and/or superficial bladder cancer.
* Symptomatic, or untreated central nervous system (CNS) lesions except stable and well controlled with no neurological symptoms; patients receiving corticosteroids to control neurological symptoms should be on stable doses for at least 14 days before study entry.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.

NOTE: Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Screening (Day ≤28) up to 28-day follow-up after end of treatment (Approximately 12 months)
  Evaluation of type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0), duration of AEs, electrocardiogram (ECG) and laboratory abnormalities

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From the date of first response up to data cut-off (approximately 12 months)
  Calculated as the proportion of evaluable patients who have achieved, as best overall response (BOR), complete response (CR) or partial response (PR) through Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Duration of response (DoR) | From the date of first response up to data cut-off (approximately 12 months)
  Duration of response will be calculated from the date of either first CR or PR until the date of documented progression for patients who achieved CR or PR. Patients who died without report of progression will be considered non-events and censored at their last disease-free assessment date
Progression-free survival (PFS) | From the date of treatment initiation up to data cut-off (approximately 12 months)
  Progression Free Survival will be calculated from the date of treatment initiation to the date of first documentation of disease progression, or death due to any cause, whichever occurs first
Overall survival (OS) | From the date of treatment initiation up to data cut-off (approximately 12 months)
  Overall Survival will be calculated from the date of treatment initiation to the date of death due to any cause
Maximum plasma concentration (Cmax) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Time to maximum plasma concentration (Tmax) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Area under the plasma concentration versus time curve up to the last detectable concentration (AUC) for NMS-03305293 | Cycle 1 - Days 1-2 and Days 5-6. Each cycle is 28 days
Minimum plasma concentration (Cmin) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Average plasma concentration (Cave) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Area under the plasma concentration versus time curve to infinity (AUCinf) for NMS-03305293 | Cycle 1 - Days 1-2 and Days 5-6. Each cycle is 28 days
Terminal elimination half-life (t1/2) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Oral plasma clearance (CL/F) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Apparent volume of distribution (Vd/F) of NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Accumulation ratio (Rac) of Cmax for NMS-03305293 | Cycle 1 - Day 1 and Day 5. Each cycle is 28 days
Rac of Area under the plasma concentration vs time curve within dosing interval (AUCdaily) for NMS-03305293 | Cycle 1 - Days 1-2 and Days 5-6. Each cycle is 28 days
Rac of Area under the plasma concentration up to the last detectable plasma concentration (AUClast) for NMS-03305293 | Cycle 1 - Days 1-2 and Days 5-6. Each cycle is 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tennessee Oncology, PLLC, Nashville, Tennessee